CLINICAL TRIAL: NCT05819957
Title: Evaluation of a Therapeutic Education Program for Multiple System Atrophy (MSA) Patients : MSA Feasibility
Brief Title: Therapeutic Education for Multiple System Atrophy (MSA) Patients and Their Caregivers
Acronym: ETP@MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/22/0520; 2023-A00340-45 (Other: ANSM)
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Multiple System Atrophy
Keywords: TherapeuticEducationProgram; Feasibility
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental patients (Experimental): MSA patients included in the therapeutic education program
  Interventions: Other: Therapeutic Education Program (TEP)

INTERVENTIONS:
Other: Therapeutic Education Program (TEP) — the TEP lasts 12 months, being structured into 6 modules.

SUMMARY:
Multiple system atrophy (MSA) is a rare neurodegenerative disorder that leads to major disability, forcing patients and caregivers to adapt their environment and lifestyle. Once they receive the diagnosis, patients and caregivers need to understand the symptoms, cope with them, to digest the diagnosis... All these needs are not completely addressed by the current model of care so we created a therapeutic educational program (TEP) program that will last 12 months, involving both patients and caregivers, including a mixed model of in-person visits and continuous on-line activities. Our project aims to target early MSA patients and their caregivers, proposing to test the feasibility (primary objective) of an innovative therapeutic educational program (TEP) for MSA patients.

DETAILED DESCRIPTION:
The announcement of MSA diagnosis may provoke a shock in patients and their relatives. Educational programs in neurodegenerative diseases, such as Parkinson's disease (PD), offer patients and caregivers structured skills in disease knowledge, expertise, and management. Those programs may result in an improvement of patients' quality of life (QoL), empowering patients and their caregivers to deal with psychosocial challenges. Additionally, it has been shown that educational programs positively impact the perceived health of PD patients without increasing medical costs. There is no educational program for MSA patients. This is the reason why we created the first therapeutic educational program (TEP) for MSA patients and caregivers, including a mix model of in person visits and online classes and virtual activities. Herein, we aim to target early MSA patients (time to diagnosis < 1 year) and their caregivers, proposing to test the feasibility of this TEP. The program will last 12 months, involving both patients and caregivers, including a mixed model of in-person visits (at baseline and 12 months) and continuous on-line activities (learning situations, questionnaires, quizzes, videos, and interactive exercises).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a clinically probable diagnosis of MSA within the last 3 years or clinically established within the last year
* Presence of a caregiver defined as a spouse, son/daughter or relative who lives with or sees the patient on a regular basis, i.e. at least three times a week.

Exclusion Criteria:

* Patients and/or caregiver unable to give consent
* Patients without access to an internet network or without the material means to access the distance learning modules
* Patients with a life expectancy of less than one year
* Patients with legal guardians, curators, or legal protection
* Patients not affiliated to a social security system
* Patients in a period of exclusion from another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the program | 1 year
  Rate of the patient/caregiver pairs having reached the visit at 6 months and the visit at 12 months of the ETP program. The threshold value of the rate being 80% = " retention rate ". Thus, if the rate is equal or above 80% : the program is considered feasable

SECONDARY OUTCOMES:
Recruitment rate | 1 year
  Rate of eligible patients successfully enrolled in the study
Satisfaction rate | 1 year
  Satisfaction of the patients and caregivers with the program will be assessed by means of Likert scale questionnaires, stratified for different aspects of the program, including content, ease of use and format. Drop-out reasons will be recorded, to better understand the needs or the difficulties met during the TEP by patients and caregivers. As routinely done for all MSA patients followed in our Reference Centres, Unified Multiple System Atrophy Rating Scale (UMSARS) I + II will be collected at baseline and at study ending (12 months) The scale goes from 0 to 10 : 10 representing the highest satisfaction of the program.

CONTACTS AND LOCATIONS:
Overall Officials: Margherita FABBRI, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France